CLINICAL TRIAL: NCT05084651
Title: A Phase I, Open-label, Fixed Sequence, Two-period, Crossover, Drug-drug Interaction Study to Investigate the Interaction Potential of Itraconazole on the Pharmacokinetics of Ganaplacide and Lumefantrine Combination in Healthy Participants
Brief Title: Drug-drug Interaction Study of Ganaplacide and Lumefantrine With Itraconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CKAF156A2105; 2021-000924-36 (EudraCT Number)
Record Dates: First submitted 2021-10-06; First posted 2021-10-20 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Malaria
Keywords: Drug-drug interaction; DDI; ganaplacide; lumefantrine; itraconazole; Cytochrome P450; CYP; Pharmacokinetic; PK; safety and tolerability; healthy participants
MeSH Terms: conditions — Malaria | interventions — ganaplacide; Lumefantrine; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): Each participant will receive a single oral dose of ganaplacide and lumefantrine combination on Day 1 of Period 1. In Period 2, participants will receive itraconazole q.d. on Days 1 to 18 and a single dose of ganaplacide and lumefantrine combination on Day 5, approximately 2 hours after the itraconazole dose
  Interventions: Drug: Ganaplacide; Combination Product: Lumefantrine; Drug: Itraconazole

INTERVENTIONS:
Drug: Ganaplacide — Treatment A/Period 1: 400 mg (4 x 100 mg tablets) at Hour 0 on Day 1 Treatment B/Period 2: 400 mg (4 x 100 mg tablets) at Hour 0, approximately 2 hours after itraconazole dosing, on Day 5.
  Other Names: KAF156
Combination Product: Lumefantrine — Treatment A/Period 1: 480 mg (2 x 240 mg sachets) at Hour 0 on Day 1 Treatment B/Period 2: 480 mg (2 x 240 mg sachets) at Hour 0, approximately 2 hours after itraconazole dosing, on Day 5.
  Other Names: LUM566
Drug: Itraconazole — 200 mg (20 mL of 10 mg/mL oral solution) q.d. on Days 1 to 18

SUMMARY:
The study will assess the effect of multiple doses of itraconazole, a strong CYP3A4/5 inhibitor, on the PK of ganaplacide and lumefantrine in healthy participants. This study will provide data that is relevant for advice regarding possible concomitant medications that are inhibitors of CYP3A4/5 in future clinical studies with ganaplacide and lumefantrine and for potential future labeling considerations

DETAILED DESCRIPTION:
This is an open-label, fixed sequence, 2-period, crossover, drug-drug interaction (DDI) study, to evaluate the effect of multiple doses of itraconazole on the single dose PK of ganaplacide and lumefantrine in healthy participants.

The study will consist of a screening period of up to 28 days, 2 Baseline evaluations (on Day -1 of each treatment period), and 2 treatment periods which are separated by a washout period. Participants who meet the eligibility criteria at Screening will be admitted to the study site for First Baseline evaluations on Day -1 of Period 1. Baseline safety assessments will be performed prior to first dosing of study treatment in each period.

Participants enrolled will receive a single oral dose of ganaplacide and lumefantrine combination on Day 1 of Period 1. In Period 2, participants will receive itraconazole once daily (q.d.) on Days 1 to 18 and a single dose of ganaplacide and lumefantrine combination on Day 5, approximately 2 hours after the itraconazole dose. There will be 336 hours of sequential blood sampling for PK assessment starting after ganaplacide and lumefantrine dosing in each treatment period. Between the 2 treatment periods, there will be an additional washout period of at least 14 days, beginning from the last PK sample collection in Period 1 and continuing until the first dose of study treatment in Period 2.

Each dose of ganaplacide and lumefantrine combination will be administered after at least 10 hours of overnight fasting and will be followed by at least 4 hours of fasting post dose. In Period 2, itraconazole will be administered after at least 10 hours of overnight fasting and followed by at least 1 hour of fasting post dose (except on Day 5 when ganaplacide and lumefantrine will be administered approximately 2 hours after itraconazole dosing and participants will continue fasting for at least 4 hours post ganaplacide and lumefantrine dosing).

Safety assessments (including physical examinations, electrocardiograms (ECGs), vital signs, clinical laboratory evaluations [hematology, chemistry, coagulation, and urinalysis], and adverse event [AE] and serious adverse event [SAE] monitoring) will be performed during the study.

The Study Completion evaluations will occur on Day 19 of Period 2, followed by a post study safety contact (e.g. follow-up telephone call, email) approximately 30 days after the last dose of study treatment. In the case of early termination, Study Completion evaluations will be conducted prior to discharge from the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Healthy male and non-childbearing potential female participants 18 to 55 years of age inclusive, at Screening.
* In good health as determined by medical history, physical examination, vital signs, ECG, and clinical laboratory tests at Screening.
* Must weigh at least 50 kg with a body mass index (BMI) within the range of 18 to 29.9 kg/m2 inclusive, at Screening.

Key Exclusion Criteria:

* Use of other investigational drugs within 5 half-lives or 30 days prior to first dosing of study treatment, whichever is longer.
* Known family history or known presence of long QT syndrome.
* Known history or current clinically significant arrhythmias.
* History or presence of malignancy of any organ system (other than treated localized basal cell or squamous cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within 5 years of Screening, regardless of whether there is evidence of local recurrence or metastases.
* History or presence of duodenal ulcer, ulcerative colitis, or Crohn's disease.
* Presence of active or uncontrolled thyroid disease.
* Has had cholecystectomy (gallbladder removed).

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-14 (Actual)

PRIMARY OUTCOMES:
Observed maximum plasma concentration (Cmax) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUCinf will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) to the 24-hour time point (AUC^0-24) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC^0-24 will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Apparent total body clearance of drug from plasma following extravascular administration (CL/F) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. CL/F will be listed and summarized using descriptive statistics.
Apparent volume of distribution during terminal elimination phase following extravascular administration (Vz/F) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Vz/F will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T^1/2) for Ganaplacide and Lumefantrine | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. T^1/2 will be listed and summarized using descriptive statistics.

SECONDARY OUTCOMES:
Observed maximum plasma concentration (Cmax) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Cmax will be listed and summarized using descriptive statistics.
Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUClast will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUCinf will be listed and summarized using descriptive statistics.
Area under the concentration-time curve from time zero (pre-dose) to the 24-hour time point (AUC0-24) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. AUC^0-24 will be listed and summarized using descriptive statistics.
Time of maximum observed drug concentration occurrence (Tmax) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. Tmax will be listed and summarized using descriptive statistics.
Terminal elimination half-life (T^1/2) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. T^1/2 will be listed and summarized using descriptive statistics.
Metabolite to Parent Ratio (MR) for Ganaplacide metabolites (RHF218 and GOU089) | 0 (pre-dose), 0.5, 1, 3, 6, 8, 12, 24, 48, 72, 96, 120, 144, 168, 240, and 336 hours (post dose)
  Venous whole blood samples will be collected for activity-based pharmacokinetics characterization. MR will be listed and summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No